CLINICAL TRIAL: NCT02741596
Title: HELP Study ExtensionTM: An Open-Label Study to Evaluate the Long-Term Safety and Efficacy of DX-2930 for Prevention Against Acute Attacks of Hereditary Angioedema (HAE)
Brief Title: Long-term Safety and Efficacy Study of DX-2930 (SHP643) to Prevent Acute Angioedema Attacks in Patients With Type I and Type II HAE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DX-2930-04; 2015-005255-27 (EudraCT Number)
Record Dates: First submitted 2016-04-08; First posted 2016-04-18 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: DX-2930(SHP643); Dyax; Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rollover Participants (Experimental): Participants who rollover from the DX-2930-03 study will receive 300 milligram (mg) DX-2930 subcutaneous injection at Day 0 followed by second dose following the first HAE attack and then once in every 2 weeks until the end of the treatment period (up to 924 days). A wash-out period of a minimum of 10 days and a maximum of 18 days is required between subsequent administrations.
  Interventions: Drug: DX-2930
- Non-rollover Participants (Experimental): Participants who were not participants in DX-2930-03 will receive 300 milligram (mg) DX-2930 subcutaneous injection once in every 2 weeks until the end of the treatment period (up to 924 days).
  Interventions: Drug: DX-2930

INTERVENTIONS:
Drug: DX-2930 — Participants who rollover from the DX-2930-03 study will receive 300 milligram (mg) DX-2930 subcutaneous injection at Day 0 followed by second dose following the first HAE attack and then once in every 2 weeks until the end of the treatment period (up to 924 days). A wash-out period of a minimum of 10 days and a maximum of 18 days is required between subsequent administrations.
  Arms: Rollover Participants
Drug: DX-2930 — Participants who were not participants in DX-2930-03 will receive 300 milligram (mg) DX-2930 subcutaneous injection once in every 2 weeks until the end of the treatment period (up to 924 days).
  Arms: Non-rollover Participants

SUMMARY:
This study is an open-label, long term safety and efficacy study to evaluate DX-2930 in preventing acute angioedema attacks in participants with Type I and Type II HAE.

ELIGIBILITY:
Inclusion Criteria:

* Male and female HAE participants who are 12 years of age or older at the time of screening
* Documented diagnosis of HAE (Type I or II) based on

  1. Documented clinical history consistent with HAE (subcutaneous or mucosal, nonpruritic swelling episodes without accompanying urticaria).
  2. Diagnostic testing results obtained during screening (or a prior DX-2930 study) that confirm HAE Type I or II: C1 inhibitor (C1-INH) functional level less than (<) 40 percentage (%) of the normal level. Participants with functional C1-INH level 40-50% of the normal level may be enrolled if they also have a C4 level below the normal range. Participants may be retested if results are incongruent with clinical history or believed by the investigator to be confounded by long-term prophylactic (LTP) use. (It is understood that C1-INH therapy may alter the lab results of C1-INH assessments; therefore, the investigator's discretion in collaboration with Medical Monitor is advised for proper documentation of eligibility).
  3. At least one of the following: Age at reported onset of first angioedema symptoms less than or equal to (<=) 30 years, a family history consistent with HAE Type I or II, or C1q within normal range.
* A historical baseline HAE attack rate of at least 1 attack per 12 weeks
* Adult participants and caregivers of participants under the age of 18 are willing and able to read, understand, and sign an informed consent form. Participants age 12 to 17, whose caregiver has provided informed consent, are willing and able to read, understand and sign an assent form.
* Males and females who are fertile and sexually active must adhere to contraception requirements for the duration of the study as

  1. Females (NOTE: Female rollover participants (those who previously participated in Study DX-2930-03 [NCT02586805]) of childbearing potential may continue to use the birth control method used during Study DX-2930-03 (NCT02586805).) of childbearing potential must agree to be abstinent or it is recommended to use highly effective forms of contraception from the screening period through 30 days after the final study visit. This includes stable doses (for 3 months prior to study screening) of combined estrogen and progestin-containing hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), progestin-only hormonal contraception associated with inhibition of ovulation, intra-uterine device (IUD, all types) or intrauterine hormone releasing systems (IUS). Notes: 1) A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception. 2) Use of a male condom with or without spermicide or cervical cap, diaphragm or sponge with spermicide or a combination (double barrier methods) are not considered highly effective.
  2. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
  3. Males, including males who are surgically sterile (post vasectomy), with female partners of childbearing potential must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final study visit.

Exclusion Criteria:

* Discontinued from DX-2930-03 (NCT02586805) after enrollment for any reason.
* If rolling over from DX-2930-03 (NCT02586805), presence of important safety concerns that would preclude participation in this study.
* Concomitant diagnosis of another form of chronic, recurrent angioedema, such as acquired angioedema (AAE), HAE with normal C1 inhibitor (also known as HAE Type III), idiopathic angioedema, or recurrent angioedema associated with urticaria.
* Dosing with an investigational drug (not including DX-2930 or other HAE therapies) or exposure to an investigational device within 4 weeks prior to screening.
* Exposure to angiotensin-converting enzyme (ACE) inhibitors within 4 weeks prior to screening or any newly initiated or dose modification of estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) 3 months prior to the screening visit.
* Unwilling to discontinue use of long-term prophylactic therapy for HAE (C1-INH, attenuated androgens, or anti-fibrinolytics) within 3 weeks after starting DX-2930 treatment.
* Any of the following liver function test abnormalities: alanine aminotransferase (ALT) > 3x upper limit of normal, or aspartate aminotransferase (AST) > 3x upper limit of normal, or total bilirubin > 2x upper limit of normal (unless the bilirubin elevation is a result of Gilbert's Syndrome).
* Pregnancy or breastfeeding.
* Participant has any condition that, in the opinion of the investigator or Sponsor, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (eg, history of substance abuse or dependence, a significant pre-existing illness or other major comorbidity that the investigator considers may confound the interpretation of study results).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (43):
- United States (31):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Institute Asthma and Allergy, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Midwest Immunology Clinic, Plymouth, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hudson-Essex Allergy, LLC, Belleville, New Jersey
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Clinical Research Center of Charlotte, Charlotte, North Carolina
  - Duke Asthma, Allergy, and Airway Center, Durham, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Optimed Research, LTD., Columbus, Ohio
  - Toledo Institute of Clinical REsearch, Toledo, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Austin Regional Clinic, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Allergy Associates of Utah, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Premier Clinical Research, Spokane, Washington
  - Medical College of Wisconsin, Childrens Hospital, Milwaukee, Wisconsin
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Yang Medicine, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Inc., Toronto, Ontario
  - Clinique Spécialisée en Allergie de la Capitale, Québec, Quebec
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Hautklinik der Universitätsmedizin Mainz, Mainz
  - HZRM Hamophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- University of Milan Luigi Sacco Hospital, Milan, Italy
- Triumpharma Clinical Evaluation Centre, Amman, Jordan
- Adler Medical Plaza, San Juan, Puerto Rico
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Craig T, Tachdjian R, Bernstein JA, Anderson J, Nurse C, Watt M, Yu M, Juethner S. Long-term prevention of hereditary angioedema attacks with lanadelumab in adolescents. Ann Allergy Asthma Immunol. 2024 Dec;133(6):712-719.e1. doi: 10.1016/j.anai.2024.08.001. Epub 2024 Aug 10. PMID 39128590
- [Derived] Lumry WR, Maurer M, Weller K, Riedl MA, Watt M, Yu M, Devercelli G, Meunier J, Banerji A; HELP OLE Study Group. Long-term lanadelumab treatment improves health-related quality of life in patients with hereditary angioedema. Ann Allergy Asthma Immunol. 2023 Jul;131(1):101-108.e3. doi: 10.1016/j.anai.2023.03.028. Epub 2023 Apr 5. PMID 37028510
- [Derived] Craig TJ, Zaragoza-Urdaz RH, Li HH, Yu M, Ren H, Juethner S, Anderson J; HELP and HELP OLE Study Investigators. Effectiveness and safety of lanadelumab in ethnic and racial minority subgroups of patients with hereditary angioedema: results from phase 3 studies. Allergy Asthma Clin Immunol. 2022 Sep 24;18(1):85. doi: 10.1186/s13223-022-00721-y. PMID 36153561
- [Derived] Banerji A, Bernstein JA, Johnston DT, Lumry WR, Magerl M, Maurer M, Martinez-Saguer I, Zanichelli A, Hao J, Inhaber N, Yu M, Riedl MA; HELP OLE Investigators. Long-term prevention of hereditary angioedema attacks with lanadelumab: The HELP OLE Study. Allergy. 2022 Mar;77(3):979-990. doi: 10.1111/all.15011. Epub 2021 Aug 13. PMID 34287942
- [Derived] Riedl MA, Bernstein JA, Craig T, Banerji A, Magerl M, Cicardi M, Longhurst HJ, Shennak MM, Yang WH, Schranz J, Baptista J, Busse PJ. An open-label study to evaluate the long-term safety and efficacy of lanadelumab for prevention of attacks in hereditary angioedema: design of the HELP study extension. Clin Transl Allergy. 2017 Oct 6;7:36. doi: 10.1186/s13601-017-0172-9. eCollection 2017. PMID 29043014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 43 sites across United States, Canada, Europe and Jorden between 26 May 2016 (first participant first visit) and 31 October 2019 (last participant last visit).
Pre-assignment Details: A total of 212 participants were enrolled and received treatment in two groups (Rollover participants [109] and Non-rollover participants [103]). Participants who rolled from the DX-2930-03 (NCT02586805) study were in Rollover group and participants who were directly enrolled into this DX-2930-04 study were in Non-rollover group.
Groups:
- Rollover Participants: Participants who rolled from the DX-2930-03 (NCT02586805) study received 300 milligrams (mg) of DX-2930 subcutaneous (SC) injection on Day 0 followed by a second dose after participants reported their first HAE attack and continued to receive repeated SC administrations of 300 mg DX-2930 every 2 weeks (q2wks) throughout the treatment period (up to 924 days). A wash-out period of a minimum of 10 days and a maximum of 18 days were required between subsequent administrations.
- Non-rollover Participants: Participants who directly entered in to this DX-2930-04 study received 300 mg of DX-2930 SC injection on Day 0 and continued to receive SC administrations of 300 mg DX-2930 every 2 weeks throughout the treatment period (up to 924 days).
Period: Overall Study
Arm/Group | Rollover Participants | Non-rollover Participants
Started | 109 | 103
Completed | 31 | 25
Not Completed | 78 | 78
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Pregnancy | 3 | 1
Not completed — Other (Unspecified) | 0 | 3
Not completed — Subject withdrawn-Other | 17 | 4
Not completed — Subject withdrawn-to commercial product | 54 | 63

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any study drug after entering the DX-2930-04 study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rollover Participants | Non-rollover Participants | Total
Number analyzed (Participants) | 109 | 103 | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (14.74) | 39.5 (16.71) | 40.7 (15.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 68 | 143
  Male | 34 | 35 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 101 | 97 | 198
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 99 | 99 | 198
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial Participant whether or not it appeared to have a causal relationship with the treatment administered. Treatment-emergent AEs were defined as AEs with onset at the time of or following the first exposure to open-label DX-2930 in this study, or medical conditions present prior to the start of treatment but increasing in severity or relationship at the time of or following the start of treatment.
Time Frame: From start of the study up to follow-up (Day 952)
Population: Safety population included all participants who received any study drug after entering the DX-2930-04 study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 109 | 103
Participants | 105 | 101

2. Secondary Outcome: Rate of Investigator Confirmed Hereditary Angioedema (HAE) Attacks During the Treatment Period
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. The treatment period investigator-confirmed HAE attack rate was calculated for each participant as the number of investigator-confirmed HAE attacks occurring during the treatment period (regular dosing stage of the treatment period for rollover participants) divided by the number of days the participant contributed to the treatment period multiplied by 28 days. Rate of investigator-confirmed HAE attacks during the treatment period was reported.
Time Frame: Up to Day 924
Population: Safety population included all participants who received any study drug after entering the DX-2930-04 study. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Attacks per month
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 106 | 103
Attacks per month | 0.27 (0.581) | 0.22 (0.521)

3. Secondary Outcome: Rate of Investigator-Confirmed Hereditary Angioedema (HAE) Attacks Requiring Acute Treatment During the Treatment Period
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Rate of investigator-confirmed HAE attacks requiring acute treatment for each participant as the number of investigator-confirmed HAE attacks occurring during the treatment period (regular dosing stage of the treatment period for rollover participants) divided by the number of days the participant contributed to the treatment period multiplied by 28 days. Rate of investigator-confirmed HAE attacks requiring acute treatment during the treatment period was reported.
Time Frame: Up to Day 924
Population: Safety population was analyzed, which included all participants who received any study drug after entering the DX-2930-04 study. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Attacks per month
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 106 | 103
Attacks per month | 0.20 (0.430) | 0.21 (0.517)

4. Secondary Outcome: Rate of Moderate or Severe Hereditary Angioedema (HAE) Attacks During the Treatment Period
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Moderate and severe investigator-confirmed HAE attacks were the attacks that were moderate or severe as per the HAE attack assessment and reporting procedures (HAARP) defined severity. The overall severity of attack was determined by the investigator using following definitions: mild (transient or mild discomfort), moderate (mild to moderate limitation in activity), severe (marked limitation in activity). Rate of moderate or severe HAE attacks during the treatment period was reported.
Time Frame: Up to Day 924
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Attacks per month
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 106 | 103
Attacks per month | 0.21 (0.479) | 0.19 (0.512)

5. Secondary Outcome: Rate of High-Morbidity Hereditary Angioedema (HAE) Attacks During the Treatment Period
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. High-morbidity Hereditary Angioedema (HAE) attack was defined as any attack that had at least one of the following characteristics: severe, resulted in hospitalization (except hospitalization for observation lesser than [<] 24 hours), hemodynamically significant (systolic blood pressure <90 millimeter of mercury [mmHg], required intravenous hydration, or associated with syncope or near-syncope) or laryngeal edema. Number of high-morbidity HAE attacks during the treatment period was analyzed and reported using the methods for the overall number of investigator-confirmed HAE attacks with the exception of the monthly line graphs. Rate of high-morbidity HAE attacks during the treatment period was reported.
Time Frame: Up to Day 924
Population: Safety population included all participants who received any study drug after entering the DX-2930-04 study. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Attacks per month
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 106 | 103
Attacks per month | 0.03 (0.085) | 0.04 (0.103)

6. Secondary Outcome: Time to First Investigator-Confirmed Hereditary Angioedema (HAE) Attacks in Rollover Participants
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Time to first investigator-confirmed HAE attack was calculated from the time of first open-label dose to the start time of the first investigator-confirmed HAE attack. Time to the first investigator-confirmed HAE attack was analyzed and reported only in rollover safety population.
Time Frame: Up to Day 924
Population: Rollover Safety Population included subset of participants who participated in the DX-2930-03 (NCT02586805) study and received any study drug after entering the DX-2930-04 study (that is any exposure to open-label DX-2930). Here, data was not planned to be collected and analyzed for Non-rollover participants.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 109 | 0
Days | 43 [18 to 97] |

ADVERSE EVENTS:
Time Frame: From start of the study up to follow-up (Day 952)
Groups:
- Rollover: Participants who rolled from the DX-2930-03 (NCT02586805) study received 300 milligrams (mg) of DX-2930 subcutaneous (SC) injection on Day 0 followed by a second dose after participants reported their first HAE attack and continued to receive repeated SC administrations of 300 mg DX-2930 every 2 weeks (q2wks) throughout the treatment period (up to 924 days). A wash-out period of a minimum of 10 days and a maximum of 18 days were required between subsequent administrations.
- Non-Rollover: Participants who directly entered in to this DX-2930-04 study received 300 mg of DX-2930 SC injection on Day 0 and continued to receive SC administrations of 300 mg DX-2930 every 2 weeks throughout the treatment period (up to 924 days).
Arm/Group | Rollover | Non-Rollover
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/103
Serious Adverse Events (participants affected / at risk) | 12/109 | 9/103
Other Adverse Events (participants affected / at risk) | 100/109 | 96/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover (N=109) | Non-Rollover (N=103)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover (N=109) | Non-Rollover (N=103)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (20) | 16 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (29) | 10 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (13) | 9 (12)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 11 (12)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (16) | 9 (14)
Toothache (Gastrointestinal disorders) | 6 (9) | 5 (6)
Vomiting (Gastrointestinal disorders) | 7 (8) | 4 (4)
Fatigue (General disorders) | 10 (15) | 10 (12)
Injection site bruising (General disorders) | 13 (21) | 13 (72)
Injection site erythema (General disorders) | 16 (40) | 20 (103)
Injection site pain (General disorders) | 45 (736) | 55 (992)
Injection site pruritus (General disorders) | 4 (5) | 6 (14)
Injection site swelling (General disorders) | 6 (49) | 11 (26)
Peripheral swelling (General disorders) | 7 (11) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 8 (8)
Acute sinusitis (Infections and infestations) | 7 (10) | 7 (11)
Bronchitis (Infections and infestations) | 5 (7) | 8 (10)
Gastroenteritis (Infections and infestations) | 4 (5) | 11 (14)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 10 (11)
Gastrointestinal infection (Infections and infestations) | 6 (7) | 4 (4)
Influenza (Infections and infestations) | 13 (17) | 9 (10)
Otitis media (Infections and infestations) | 6 (7) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 3 (3) | 6 (8)
Sinusitis (Infections and infestations) | 13 (13) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 30 (51) | 25 (54)
Urinary tract infection (Infections and infestations) | 10 (12) | 13 (21)
Viral upper respiratory tract infection (Infections and infestations) | 51 (119) | 38 (87)
Contusion (Injury, poisoning and procedural complications) | 8 (9) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (7) | 12 (14)
Procedural pain (Injury, poisoning and procedural complications) | 7 (9) | 4 (5)
Alanine aminotransferase increased (Investigations) | 4 (9) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 6 (8)
Blood creatine phosphokinase increased (Investigations) | 7 (8) | 5 (8)
Headache (Nervous system disorders) | 29 (70) | 23 (37)
Anxiety (Psychiatric disorders) | 8 (9) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (9)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02741596/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT02741596/SAP_001.pdf